CLINICAL TRIAL: NCT00001004
Title: A Randomized Multicenter Phase II Trial of Recombinant Tumor Necrosis Factor and Recombinant Human Interferon-gamma in Patients With AIDS Related Complex
Brief Title: A Study of Tumor Necrosis Factor and Human Interferon-gamma in Patients With AIDS Related Complex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 025; 11001 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Tumor Necrosis Factor; Interferon-gamma, Recombinant; HIV Antigens; Immunologic Surveillance; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Tumor Necrosis Factor-alpha; interferon gamma-1b

INTERVENTIONS:
Drug: Tumor Necrosis Factor
Drug: Interferon gamma-1b

SUMMARY:
To study the tolerance and toxicity of the combination of tumor necrosis factor (TNF) and interferon gamma (IFN-G) or as single agent TNF or IFN-G in HIV infected patients. To selectively monitor the immune system of AIDS related complex (ARC) patients who receive either combination therapy or TNF or IFN-G alone. To obtain information on the effectiveness of combination therapy or TNF or IFN-G alone against HIV in ARC patients.

Recombinant TNF and recombinant IFN-G have been shown to be effective against the virus which causes AIDS and ARC in some laboratory studies, but may increase virus replication in other laboratory studies. Previous studies in humans showed no increase in virus cultures and some decrease in measurements of virus. Extensive preclinical data show that TNF and IFN-G are more effective together than separately in laboratory and animal studies. As single agents, both TNF and IFN-G have modest effect against HIV. Studies have demonstrated that TNF and IFN-G, in combination, can not only inhibit HIV infection of previously uninfected cells, but also can selectively induce the destruction of acutely infected target cells.

DETAILED DESCRIPTION:
Recombinant TNF and recombinant IFN-G have been shown to be effective against the virus which causes AIDS and ARC in some laboratory studies, but may increase virus replication in other laboratory studies. Previous studies in humans showed no increase in virus cultures and some decrease in measurements of virus. Extensive preclinical data show that TNF and IFN-G are more effective together than separately in laboratory and animal studies. As single agents, both TNF and IFN-G have modest effect against HIV. Studies have demonstrated that TNF and IFN-G, in combination, can not only inhibit HIV infection of previously uninfected cells, but also can selectively induce the destruction of acutely infected target cells.

Patients with ARC who are positive for HIV antibody are randomized to receive one of three treatment arms: (1) TNF alone by intramuscular injection (IM); (2) IFN-G alone by IM; (3) TNF plus IFN-G. Patients receive IM injections 3 times weekly for 4 months (16 weeks). Repeated physical examinations and laboratory tests are used to monitor patients' safety. Serial HIV cultures and core antigen assays are employed to obtain evidence of antiviral activity and serial T cell and skin tests are used to measure immunologic effect.

ELIGIBILITY:
Inclusion Criteria

Patients who have a primary diagnosis of AIDS related complex (ARC) including lymphadenopathy syndrome (LAS), who are positive for HIV antibody, have a minimum life expectancy of 3 months, and have one or more of the following symptoms for = or > 30 days:

* Fever.
* Night sweats.
* Fatigue.
* Oral thrush.
* Hairy leukoplakia.
* Diarrhea.
* Weight loss < 10 percent.
* Patients must be able to sign a written informed consent form, which must be obtained prior to treatment.

Concurrent Medication:

Allowed:

* Acetaminophen for temperature rise of > 38.5 degrees C - 650 mg by mouth every 4 hours on an as needed basis.

Severe rigors may be treated (or prevented) with meperidine 50 mg IV on an as needed basis in the absence of systolic hypotension < 80 mm Hg.

-

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Clinically significant cardiac disease - New York Heart Association Class II, III, or IV.
* Hemorrhagic diathesis (including hemophilia) or active bleeding disorder (e.g., genitourinary, gastrointestinal).
* Clinically apparent vascular disease (including a prior history of pulmonary embolus, deep venous thrombosis, or peripheral arterial occlusive disease).

Concurrent Medication:

Excluded:

* Medications required for the treatment of active cardiac disease including cardiac glycosides, antiarrhythmics and antianginal agents.
* Anticoagulants.
* Thrombolytic agents.
* Nonsteroidal anti-inflammatory drugs.
* Ongoing therapy with vasodilators.
* Aspirin.
* Corticosteroids.
* Antihistamines.
* Barbiturates.
* Excluded within 4 weeks of study entry:
* Antiviral chemotherapy.
* Immunotherapy.
* Excluded within 12 weeks of study entry:
* Suramin.

Patients with the following are excluded:

* AIDS-associated opportunistic infection.
* Lipoprotein disorders.
* Hemophilia.

Prior Medication:

Excluded:

* Interferon gamma.
* Tumor necrosis factor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaplan L, Study Chair; Corey L, Study Chair
Locations (1):
- Univ of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Agosti JM, Coombs R, Kidd PG, Paradise M, Sherwin S, Corey L. Randomized phase II trial of recombinant tumor necrosis factor (rTNF) and recombinant interferon-gamma (rIFN-gamma) in patients with ARC. Int Conf AIDS. 1989 Jun 4-9;5:558 (abstract no MCP101)
- [Background] Agosti JM, Coombs RW, Collier AC, Paradise MA, Benedetti JK, Jaffe HS, Corey L. A randomized, double-blind, phase I/II trial of tumor necrosis factor and interferon-gamma for treatment of AIDS-related complex (Protocol 025 from the AIDS Clinical Trials Group). AIDS Res Hum Retroviruses. 1992 May;8(5):581-7. doi: 10.1089/aid.1992.8.581. PMID 1515211